CLINICAL TRIAL: NCT00161876
Title: Open-label, Multicenter, Follow-up Phase III Study to Investigate the Safety of the Third Vaccination of FSME-IMMUN NEW in Volunteers Aged 16 to 66 Years
Brief Title: FSME IMMUN NEW Follow-up to Study 208 in Volunteers Aged 16 to 66 Years
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 213
Record Dates: First submitted 2005-09-08; First posted 2005-09-13 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Encephalitis, Tick-borne
Keywords: tick-borne encephalitis
MeSH Terms: conditions — Encephalitis, Tick-Borne | interventions — Vaccines

INTERVENTIONS:
Biological: Tick-Borne Encephalitis (TBE) Vaccine (Inactivated)

SUMMARY:
The aim of this study is to evaluate the safety of the third vaccination with FSME-IMMUN NEW in all volunteers who received both vaccinations in Baxter study 208 (safety study of FSME IMMUN NEW and ENCEPUR in healthy volunteers aged 16 to 65 years).

ELIGIBILITY:
Inclusion Criteria:

* Received two vaccinations during the course of Baxter study 208
* Understand the nature of the study, agree to its provisions and give written informed consent
* For volunteers under 18 years of age - written informed consent of the parents/legal guardian is given

Exclusion Criteria:

* None.

Volunteers assessed for eligibility to receive a third vaccination.

Eligibility to receive third vaccination:

* ELISA value > 126 VIE U/ml before the first TBE vaccination in Baxter study 208
* Not clinically healthy, (i.e. the physician would have reservations vaccinating with FSME-IMMUN NEW outside the scope of a clinical trial)
* Have already been administered a third TBE vaccination elsewhere since receiving the two vaccinations in Baxter study 208
* Have had an allergic reaction to one of the components of the vaccine since the last vaccination in Baxter study 208
* Suffer from a disease (e.g. autoimmune disease) or are undergoing a form of treatment (e.g. systemic corticosteroids, chemotherapeutics) that can be expected to influence immunological functions
* Have a known or suspected problem with drug or alcohol abuse (> 4 liters wine / week or equivalent dose of other alcoholic beverages)
* Have received banked human blood or immunoglobulins within one month of study entry
* Are known to have become infected with HIV (a special HIV test is not required for the purpose of the study) since the last visit of study 208
* Have had a vaccination against yellow fever and / or Japanese B-encephalitis since the last visit in study 208
* Have received an investigational new drug within 6 weeks prior to study start
* Have a positive pregnancy test at the first medical examination (for females capable of bearing children)
* Do not agree to employ adequate birth control measures for the duration of the study (for females capable of bearing children)

Ages: 16 Years to 66 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3973
Dates: Start 2002-05; Study Completion 2002-08

CONTACTS AND LOCATIONS:
Overall Officials: Jerzy Romaszko, MD, Principal Investigator — PANTAMED sp. z o o.; Jerzy Brzostek, MD, Principal Investigator — Zespol Opieki Zdrowotnej w Debicy; Jerzy Dziduch, MD, Principal Investigator — Samodzielny Publiczny Zaklad Opieki Zdrowotnej Oddzial Pediatryczny; Krystyna Jurowska, MD, Principal Investigator — Przedsiebiorstwo Uslug Medycznych "Centrum Medyczne Nowa Huta"; Marian Patrzalek, MD, Principal Investigator — Wojewodzki Szpital Dzieciecy Oddzial Obserwacyjno - Zakazny A; Krzysztof Sladek, MD, Principal Investigator — "Atopia" Diagnostyka i Leczenie Chorob Alergicznych i Ukladu Oddechowego; Ryszard Konior, Principal Investigator — Szpital Jana Pawla II Oddzial Neuoinfekcji; Grazyna Zawada-Skrobisz, MD, Principal Investigator — Oddzial Chorob Zakaznych Specjalistyczny Szpital, Tarnow
Locations (8):
- Poland (8):
  - Zespol Opieki Zdrowotnej w Debicy, Dębica
  - Wojewodzki Szpital Dzieciecy Oddzial Obserwacyjno - Zakazny A, Kielce
  - "Atopia" Diagnostyka i Leczenie Chorob Alergicznych i Ukladu Oddechowego, Krakow
  - Przedsiebiorstwo Uslug Medycznych "Centrum Medyczne Nowa Huta", Krakow
  - Szpital Jana Pawla II Oddzial Neuroinfekcji, Krakow
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej Oddzial Pediatryczny, Lubartów
  - PANTAMED sp. z o.o., Olsztyn
  - Oddzial Chorób Zakaznych Specjalistyczny Szpital im. E. Szczeklika, Tarnów